CLINICAL TRIAL: NCT06513624
Title: A Phase 1B Investigator Initiated Study To Evaluate The Preliminary Activity, Safety And Tolerability Of ETC-159 In Combination With Pembrolizumab In Advanced MSS/pMMR Ovarian Cancers.
Brief Title: ETC-159 In Combination With Pembrolizumab In Advanced MSS/pMMR Ovarian Cancers
Acronym: ETC-159-02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: EDDC (Experimental Drug Development Centre), A*STAR Research Entities (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC-159-02
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: With MSS/pMMR Advanced, Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — ETC-159; pembrolizumab; Denosumab; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Patients will undergo screening procedures to determine eligibility within 28 days prior to the initial administration of ETC-159 in combination with pembrolizumab. ETC-159 in combination with pembrolizumab will be administered in 21-day cycles (1 cycle: 21 days). ETC-159 will be dosed every other day. Pembrolizumab will be dosed IV Q3W. Tumor response assessments will be done every 6 weeks (2 cycles) prior to starting the cycle starting at C3D1 (- 7 days) until C9D1 (- 7 days); thereafter every 12 weeks (4 cycles) starting at C13D1 (- 7 days) and at EOT, until disease progression or start of another anti-cancer therapy according to RECIST v1.1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETC-159 (Experimental): Patients will undergo screening prior to the initial administration of ETC-159 in combination with pembrolizumab. ETC-159 in combination with pembrolizumab will be administered in 21-day cycles. ETC-159 will be dosed every other day while Pembrolizumab will be dosed at IV Q3W along with bone protective treatment (Denosumab or Zoledronic Acid)
  Interventions: Drug: ETC-159; Drug: Pembrolizumab; Drug: Denosumab / Zoledronic Acid

INTERVENTIONS:
Drug: ETC-159 — ETC-159 will be administered orally.
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously.
Drug: Denosumab / Zoledronic Acid — Denosumab will be administrated subcutaneously. Zoledronic Acid will be administered intravenously if denosumab has no response.

SUMMARY:
This is an open-label, single-arm, investigator-initiated study conceived as a dose expansion cohort of the study D3-002, which evaluated ETC-159 in combination with pembrolizumab in solid tumors.

DETAILED DESCRIPTION:
Hypothesis:

Wnt pathway inhibition with ETC-159 in combination PD1 checkpoint inhibition is safe and effective for the treatment of patients with advanced MSS/pMMR ovarian cancer.It is hypothesized that, ETC-159, as a selective PORCNi, will lead to increased immune infiltration and therefore may turn "cold" tumors into "hot" tumors that may then be responsive to checkpoint inhibitor

Primary Objectives:

1. To evaluate the preliminary clinical activity of ETC-159 in combination with pembrolizumab according to RECIST v1.1, in patients with advanced or metastatic, platinum-resistant MSS/pMMR ovarian cancer
2. To assess the safety of ETC-159 at the dose of 8 mg every other day (the recommended dose [RD] identified in safety segment) in combination with pembrolizumab.

Secondary Objectives:

1. To further assess the efficacy of ETC-159 in combination with pembrolizumab
2. To evaluate the PK of ETC-159 in combination with pembrolizumab in patients.

Exploratory Objectives:

1. To evaluate the effect of ETC-159 administered orally every other day in combination with pembrolizumab with bone protective treatment (denosumab and subsequently zoledronic acid if no response is observed with denosumab) on bone turnover markers as potential downstream markers of Wnt signaling (β-CTX).
2. To correlate available tumor genomic profile with clinical data.
3. To evaluate the effect of ETC-159 treatment on :

   * Pharmacodynamic biomarker (Axin2 mRNA expression levels) in hair follicles.
   * Gene expression levels and PD-L1 protein expression measured in FFPE-tumor tissue (if sufficient tissue is available).
4. To determine change in serum levels of cancer antigen 125 (CA-125).

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with the protocol requirements.
2. Is female, and age 21 years or older (Singapore sites) at pre-screening or screening.
3. Has histologically or cytologically confirmed, advanced or metastatic ovarian cancer with a platinum free interval of less than 6 months from prior platinum based treatment or for whom platinum therapy is no longer an option according to the treating physician
4. Has MSS/pMMR tumors as determined by immunohistochemistry (IHC), polymerase chain reaction (PCR), or next-generation sequencing (NGS).
5. Has objective (assessable through clinical signs, symptoms, and/or laboratory findings) and radiologically-confirmed progression of disease at Screening.
6. Has measurable disease as determined by RECIST v1.1 (Appendix 4, Section 12.4). Target lesions should not be selected in previously irradiated fields unless there is clear evidence of progression.
7. Has ECOG performance of status 0 to 2 at Screening.
8. Has life expectancy of at least 3 months at Screening.
9. Has adequate organ function at Screening, including the following (noting that repeated tests Screening should not be performed unless there are sufficient reasons to assume the patient would meet the inclusion criteria with re-testing).

   * Absolute neutrophil count ≥1.0 × 109/L
   * Platelet count ≥100 × 109/L (without transfusions within 21 days prior to Day 1 of Cycle 1
   * Hemoglobin ≥9 g/dL
   * Prothrombin time and partial thromboplastin time within ≤1.5 × upper limit of normal (ULN)
   * International normalized ratio (INR) ≤1.5 × ULN Note: If the patient is on allowed anti-coagulants the INR and coagulation parameters should be in the therapeutic range
   * Total bilirubin ≤1.5 × ULN
   * Transaminases (AST and/or alanine aminotransferase ≤2.5 × ULN (<5 × ULN if liver metastases)
   * Calculated creatinine clearance ≥40 mL/min (Cockroft and Gault formula)
   * Total calcium (corrected for serum albumin) within normal limits prior to Day 1 of Cycle 1 (supplementation is permitted).

   Note: Patients with grade 1 changes can be included as long as they are asymptomatic and can receive supplementation during the study.

   o Magnesium ≥the lower limit of normal (LLN) prior to Day 1 of Cycle 1 (supplementation is permitted).

   Note: Patients with grade 1 changes can be included as long as they are asymptomatic and can receive supplementation during the study.
10. Patients must have a T-score greater than -1 to be eligible, however, patients with osteopenia (defined as a T-score of -1 to -2.5 at the left or right total hip, left or right femoral neck, or lumbar spine [L1 to L4] as determined by DEXA at Screening) are eligible to participate and will receive calcium and vitamin D supplements during the study. Patients with osteoporosis (T-score of <-2.5) must be excluded.

    Note: T-score should be calculated according to local requirements by DEXA scan for the purpose of determining eligibility.
11. Is capable of swallowing study medication and following directions regarding taking study drug or has a daily caregiver who will be responsible for administering study drug.
12. Has a negative serum pregnancy test at Screening or a negative urine pregnancy test within 7 days prior to Day 1 Cycle 1 prior of treatment (applies to females of childbearing potential only).
13. For all patients: pre-dose and post-dose tumor biopsies are mandatory unless tumor is inaccessible or deemed unsafe for procedure by the principal investigator.

Note: NGS reports can be collected where biopsies are not done.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

Patients meeting any of the following criteria will be excluded from the study (note that exclusion criteria must be assessed at the Screening Visit, unless otherwise specified):

1. Has received anti-cancer therapy including immunotherapy within 4 weeks (28 days) prior to starting study drug or the side effects of such therapy have not resolved to Grade ≤1 within 4 weeks prior to starting study drug or is receiving any concomitant anti-cancer therapy.
2. Has used other investigational drugs within 4 weeks (28 days) or five half-lives (whichever is longer) prior to the first dose of study drug.
3. Has evidence of another malignancy not in remission or history of such a malignancy within the last 3 years (except for treated basal or squamous cell carcinoma of the skin, or in situ cancer of the cervix).
4. Has central nervous system metastases, unless previously treated with surgery, whole-brain radiation or stereotactic radiosurgery, and stable disease for at least 8 weeks without steroid use for at least 4 weeks (28 days) prior to the first dose of ETC-159.
5. Has received prior radiation therapy within 4 weeks (28 days), or limited field radiation within 2 weeks, prior to starting study drug, or the side effects of such therapy have not resolved to Grade ≤1.
6. Has any history of direct radiation to spine or pelvis bone or definitive chemoradiation to pelvic organs in the last 6 months prior to starting study drug, or the side effects of such therapy have not resolved to Grade ≤1.
7. Has a history of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity, or pneumonitis.
8. Has received bisphosphonate therapy for osteoporosis or symptomatic hypercalcemia or denosumab for osteoporosis within 6 months prior to starting study drug.
9. Has osteoporosis based on a T-score of < -2.5 at the left or right total hip, left or right femoral neck, or lumbar spine (L1 to L4) as determined by DEXA scan at Screening (for details of calculating T-score for eligibility see Inclusion Criterion 10).
10. Has a history of symptomatic vertebral fragility fractures or any fragility fracture of the hip, pelvis, wrist, or other location (a fragility fracture is defined as any fracture without a history of trauma or as a result of a fall from standing height or less).
11. Has moderate (25% to 40% decrease in the height of any vertebra) or severe (>40% decrease in the height of any vertebra) morphometric vertebral fractures at Screening.
12. Has a β-CTX serum level >1000 pg/mL in the morning after at least 10 hours of fasting at Screening.

    Note: Patients should begin their treatment with the bone protective treatment (denosumab with a starting dose of 120 mg, administered SC), and continued so as to have a β-CTX serum level ≤1000 pg/mL
13. Has thyrotropin level less than LLN at Screening
14. Has 25-hydroxy vitamin D levels less than 25 nmol/L (10 ng/mL) at screening. Note: For patients known to have less than 25 nmol/L (10 ng/mL) 25-hydroxy vitamin D value that would otherwise be eligible to participate in the study, a single administration of oral vitamin D3 (cholecalciferol) of 100,000 IU or 2 × 50,000 IU is recommended. After a single large dose of vitamin D3, the 25-hydroxy vitamin D level is expected to return to the required range within 7 to 28 days. After the documentation of 25-hydroxy vitamin D level normalization, maintenance treatment can be started by means of oral administration of 1000 IU/day of vitamin D3 or higher, based on the investigator's clinical judgement. While vitamin D3 (cholecalciferol) is recommended for 25-hydroxy vitamin D level restoration and maintenance, equivalent doses of vitamin D2 (ergocalciferol) can be used if vitamin D3 is not available.
15. Has bone metastases at Screening.
16. Has a metabolic bone disease, such as hyperparathyroidism, Paget's disease, or osteomalacia.
17. Cannot start treatment with the bone protective treatment with denosumab and/or zoledronic acid. Cannot start treatment with the bone protective treatment with denosumab SC, in patients requiring this treatment at the start of study.
18. Is receiving active treatment with an oral or IV glucocorticoid for ≥4 weeks (≥28 days) at a daily dose equivalent to ≥10 mg of oral prednisone within the 12 weeks prior to starting the ETC-159.
19. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy [less than 10 mg prednisone or equivalent daily] for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
20. Is a female patient of childbearing potential, defined as a female physiologically capable of becoming pregnant (including a female whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, and females whose partners have been sterilized by vasectomy or other means), unless they are using a highly effective method for birth control throughout the study and for 12 weeks after the EOT. Highly effective methods for birth control include the following:

    * Total abstinence: This is an acceptable method when this is consistent with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization: The patient has had a surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks prior to taking study drug. In case of an oophorectomy alone, the reproductive status of the patient must have been confirmed by follow-up hormone level assessment.
    * Male partner sterilization: The patient has the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. (For female patients on the study, the vasectomized male partner should be the sole partner for that patient.) These patients must also agree to the following:

      * Use of a combination of the following (1+2):

        * Placement of an intrauterine device or intrauterine system
        * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, or cream, or vaginal suppository
      * Reliable contraception maintained throughout the study and for 12 weeks after study drug discontinuation
    * Females considered post-menopausal and not of childbearing potential: The definition applies to females who have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks prior to starting treatment. In the case of oophorectomy alone, only when the reproductive status of the patient has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
21. Is a pregnant or nursing (lactating) female, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test (>5 mIU/mL).
22. Has had a major surgical procedure within 4 weeks (28 days) from starting the study drug. Patient has not fully recovered from all surgery-related complications to Grade ≤1.
23. Has a history of long QT syndrome or prolonged QT interval corrected (QTc) (>460 ms) at Screening. Both Bazett's and Fridericia's QTc are accepted and should be used consistently through the study (either Bazett's or Fridericia's QTc).
24. Has a known clinically significant bleeding disorder or coagulopathy.
25. Is receiving or has received within 4 weeks prior to starting study drug, heparin, warfarin, or other similar anti-coagulants, except for patients on low molecular weight heparin or Direct-Acting Oral Anticoagulants (DOACs: factor Xa or direct thrombin inhibitors) for treatment or prophylaxis.
26. Has severe or unstable medical conditions such as heart failure, ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, an ongoing cardiac arrhythmia requiring medication (Grade ≥2, according to National Cancer Institute [NCI] CTCAE Version 4.03), or any other significant or unstable concurrent medical illness that in the opinion of the investigator would preclude protocol therapy.
27. Has a known history of human immunodeficiency virus, or active infection with hepatitis B (unless DNA count < 500) or hepatitis C virus or other active bacterial, viral, or fungal infections.
28. Has a history of gastric bypass surgery.
29. Has a serious non-healing wound, or vasculitis.
30. Has received prior treatment with an inhibitor of the Wnt-β-catenin pathway other than the study drug in question or received wnt-immunotherapy combinations.
31. Is unwilling to or unable to comply with the protocol.
32. Patient is unable to provide tumor tissue unless approved by the lead- sponsor investigator
33. Has received prophylactic administration of hematopoietic colony stimulating factors (colony stimulating factors, e.g., granulocyte colony stimulating factor, granulocyte/macrophage colony stimulating factor, pegfilgrastim, epoetin, darbepoetin) within 4 weeks (28 days) prior to starting study drug.
34. Has recent or current active infectious disease requiring systemic antibiotics or antifungal or antiviral treatment within 2 weeks (14 days) prior to the start of study drug. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible.
35. Has received a live vaccine within 28 days prior to the start of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines with attenuated live virus for injection are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are not allowed. Anti-SARS-CoV-2 live virus vaccines developed that utilized a replication-deficient simian adenoviral vector (ChAdOx1) should be avoided.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Is female, and age 21 years or older (Singapore sites) at pre-screening or screening.
Enrollment: 16 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 1 Year
  is defined as percentage of subjects with best overall response as (Complete Response (CR) + Partial Response (PR) + Stable disease ≥12 weeks) evaluated by RECIST v1.1 criteria measured by CT or MRI
Objective Response Rate (ORR) | 1 Year
  is defined as percentage of subjects with best overall response as (Complete Response (CR) + Partial Response (PR)) evaluated by RECIST v1.1 criteria measured by CT or MRI

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Pan S, Hsieh MH, Ng N, Sun F, Wang T, Kasibhatla S, Schuller AG, Li AG, Cheng D, Li J, Tompkins C, Pferdekamper A, Steffy A, Cheng J, Kowal C, Phung V, Guo G, Wang Y, Graham MP, Flynn S, Brenner JC, Li C, Villarroel MC, Schultz PG, Wu X, McNamara P, Sellers WR, Petruzzelli L, Boral AL, Seidel HM, McLaughlin ME, Che J, Carey TE, Vanasse G, Harris JL. Targeting Wnt-driven cancer through the inhibition of Porcupine by LGK974. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20224-9. doi: 10.1073/pnas.1314239110. Epub 2013 Nov 25. PMID 24277854
- [Background] DeVito NC, Sturdivant M, Thievanthiran B, Xiao C, Plebanek MP, Salama AKS, Beasley GM, Holtzhausen A, Novotny-Diermayr V, Strickler JH, Hanks BA. Pharmacological Wnt ligand inhibition overcomes key tumor-mediated resistance pathways to anti-PD-1 immunotherapy. Cell Rep. 2021 May 4;35(5):109071. doi: 10.1016/j.celrep.2021.109071. PMID 33951424